CLINICAL TRIAL: NCT03025516
Title: Performance Evaluation of Two Diagnostic Technologies for TB Detection Based Upon Breath Testing
Brief Title: Performance Evaluation of TB Breath- and Cough-testing Platforms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Find (Other)
Collaborators: Universidad Peruana Cayetano Heredia (Other); University of Cape Town (Other)
Responsible Party: Sponsor
Other Study IDs: P07212-00
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary TB; Diagnoses Diseases
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All consenting patients are expected to provide the following samples: 2x breath/cough samples, which will be collected directly into enclosed diagnostic devices and destroyed immediately following diagnosis; blood samples for HIV testing, which will be de-identified and stored until study completion; urine samples; and 3x sputum samples, collected at enrollment and during an 8-week follow-up, de-identified and used for liquid culture, solid culture, AFB smear, and DNA extraction for Xpert testing. Except for the breath samples, all samples will be de-identified and stored until study completion.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults with pulmonary TB symptoms: All patients will be tested with both the reference and index TB diagnostic tests. Index test results will not be used to inform case management.
  All samples must be collected before the patient starts any form of TB treatment. Patients will be randomized to receive either the TB Breathalyser or AeonoseTM on Day 1, and will be tested with the remaining breath-test on Day 2. A follow-up evaluation will be required after 8 weeks for all patients who do not have microbiologic confirmation of TB (smear or culture). Two additional breath samples may also be collected upon follow-up.
  Interventions: Device: Rapid Biosensor Systems (RBS) TB Breathalyser; Device: eNose AeonoseTM

INTERVENTIONS:
Device: Rapid Biosensor Systems (RBS) TB Breathalyser — Rapid Biosensor Systems (RBS) recently developed a portable, non-invasive, rapid TB diagnostic 'Breathalyser' capable of diagnosing TB in patient breath samples collected while patients cough (Figure 1). The TB Breathalyser comprises a disposable, single-use sample collection tube and a multi-use reader. At the bottom of the collection tube is a glass bio-sensor coated with a biochemical sensor that is formulated to react with TB bacilli. Patients cough into the collection tube after nebulization with 0.9% saline solution. Following sample collection, the tube is placed into the reader, where a diode laser interrogates the biochemical coating in the sample collection tube and reports the presence of TB bacilli. The entire process takes about two minutes.
Device: eNose AeonoseTM — The eNose Company has also developed a hand-held, non-invasive rapid TB diagnostic 'electronic nose' (AeonoseTM) for TB detection based upon analysis of exhaled breath. After the device has been calibrated, the patient is instructed to breathe into the device through a mouthpiece for 5 minutes. Within the device is a micro-hotplate, metal-oxide sensor which behaves as a semiconductor at high temperature. Redox-reactions occurring at the sensor surface result in changes in resistance, with results read and interpreted by a phone application to confirm the presence of MTB.

SUMMARY:
This will be a prospective, multicentre study conducted to evaluate the diagnostic accuracy of two TB breath-based technologies independently of the manufacturers. Assay error and failure rates and device operational characteristics will also be assessed during this study. Participants will be enrolled in this study in line with FIND sample banking activities. Results from index tests will not be used to make clinical decisions. Participation in this study will not alter the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms suggesting pulmonary TB, i.e. persistent cough (generally > 3 weeks or as per local definition of TB suspect) and at least one other finding listed below:

  1. Persistent cough
  2. Fever
  3. Malaise
  4. Recent weight loss
  5. Night sweats
  6. Contact w/ active case
  7. Hemoptysis
  8. Chest pain
  9. Loss of appetite
  10. Other [specify]
* Provision of informed consent to sample collection, banking and HIV and breath-based assay testing
* Production of adequate quantity of sputum (sputum induction whenever possible)
* Adult age (>18 years old)

Exclusion Criteria:

* Participants receiving any anti-tuberculosis medication, including fluoroquinolone and aminoglycosides in the 60 days prior to enrolment.
* Participants with ONLY extra-pulmonary disease will be excluded.
* Participants for whom complete follow-up and a clear final diagnosis are judged to be difficult (e.g. residents elsewhere or about to move).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult patients who have symptoms consistent with pulmonary TB presenting to health facilities during study period. Patients will be asked by study or non-study clinicians or staff if they would be interested in participating in the study. Interested individuals will be referred to study personnel for additional information and screening, if appropriate, samples will be obtained following the informed consent process.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2017-05-29 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Microbiological TB Diagnosis | 8 weeks
  TB diagnosed by AFB smear microscopy or by one of two MGIT (liquid) or LJ (solid) cultures on enrollment or follow-up sputum sample

CONTACTS AND LOCATIONS:
Overall Officials: Timothy C Rodwell, MD, PhD, MPH, Study Director — Find
Locations (1):
- Nolungile Clinic, University of Cape Town, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No